CLINICAL TRIAL: NCT02190097
Title: PALEOLITHIC VS Healthy ADA DIETS FOR TREATMENT OF POLYCYSTIC OVARIAN SYNDROME (PCOS)
Brief Title: Paleo Versus Healthy ADA Diets for Treatment of Polycystic Ovarian Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-13770
Record Dates: First submitted 2014-06-20; First posted 2014-07-15 (Estimated); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Polycystic Ovarian Syndrome
Keywords: PCOS; insulin sensitivity; paleolithic diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Diet, Paleolithic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- paleolithic diet (Experimental): subjects in this arm are given detailed instructions and coaching in following a paleolithic type diet for 4 months, with the option to continue for another 4 months. studies of ovarian and metabolic parameters will be done at baseline, 2 and 4 months
  Interventions: Other: Paleolithic diet
- American Diabetes Association diet (Active Comparator): subjects in this arm are given detailed instructions and coaching in following an ADA type diet for 4 months, with the option to switch over to the paleolithic diet arm for another 4 months. studies of ovarian and metabolic parameters will be done at baseline, 2 and 4 months
  Interventions: Other: American Diabetes Association diet

INTERVENTIONS:
Other: Paleolithic diet — see procedures section for more details
  Arms: paleolithic diet
Other: American Diabetes Association diet — see procedures section
  Arms: American Diabetes Association diet

SUMMARY:
Polycystic ovary syndrome (PCOS) is a syndrome which includes elevated androgen levels, irregular menstrual cycles and insulin resistance. Standard treatments, which include weight loss and medications to improve insulin secretion are only partly successful, and may require that young women take medications for decades.

The study investigators have been evaluating the effects of specific diets on insulin resistance in healthy volunteers and subjects with type 2 diabetes, and have found that subjects with insulin resistance seem to respond particularly well to these diet regimens.

Volunteers with PCOS are being asked to participate to see if following these diets can help regularize your menstrual cycles. The results of this study may help improve fertility treatments for women with PCOS.

DETAILED DESCRIPTION:
Experimental Design and Methods This is a prospective, open labeled, randomized diet intervention study done on adult participants with PCOS. After signing informed consents, participants will be asked to eat a recommended ADA diet for two weeks (run in period). Participants will then have baseline testing, including: urine and blood tests to evaluate insulin resistance (fasting glucose and insulin, 2 hour oral glucose tolerance test), electrolytes to assess acid-base status, ovarian volume and testosterone levels measured to assess severity of PCOS, and questionnaires about menstrual frequency, eating habits and stress. Participants will then be randomized to either a high fruits and vegetable Paleo Diet for 4-8 months or a standard ADA-recommended diet for the first 4 months followed by Paleo Diet for 0-4 months.All participants will have the option of limiting their participation to just 4 months or extending participation to the full 8 months depending on their ongoing level of interest. All testing will be repeated at 4 months (crossover point) and at completion of the diets at 8 months. The primary outcome variables are menstrual cycle frequency and ovarian volume, and secondary outcomes include metabolic profiles and eating/behavior questionnaires

Procedures

1. Diet: All participants will initially be given diet information on ADA diet for the "Run In" period , including printed ADA diet instructions and advice on caloric intake. The ADA diet includes foods that are excluded in the Paleo Diet, such as grains, legumes and dairy products and will also contain less potassium. All participants will be instructed not to add salt to their food when cooking or eating. At 2 weeks, participants will be randomized to Paleo Diet arm or ADA diet arm. Participants on the Paleo Diet arm will require a "ramp-up" phase for one week (start out with 1 Paleo meal per day, then two, and then all meals will be on a Paleolithic-type menu, which contains approximately an average of 142 grams of protein and 12,200 mg of potassium per 3000 kcal. Participants on the ADA diet arm will continue on the run-in diet.

   After 16 weeks, the participants in the ADA arm will be changed over to the Paleo arm if they wish to continue participation. They will also require a "ramp-up" phase for 1 week. In our previous studies, we have seen a crossover effect at one month going from the Paleo to the ADA diet, but not from the ADA to the Paleo arm.

   We will give all participants pertinent websites and written information about their specific diet, as well as sample menus. We will give participants in the Paleo arm a list of foods to avoid (e.g., dairy, grains, legumes, processed foods).

   The main obstacles to compliance with outpatient diets include the cost, the amount of time needed, and ignorance about where to get specific kinds of foods. We will give them lists of various supermarkets and farmers markets times and dates, we will advise participants about making up batches of foods on the weekends and freezing them, and if they have families or other support, we will try to get them involved in support.
2. Monitoring dietary compliance: We will monitor compliance in a number of ways.

We have recruited four nutrition student volunteers from UC Berkeley, who will work closely with the participants to help them adapt the study diets to their everyday living situations. The nutrition students will help design the materials we will give the participants, as well as give dietary advice. We are working on a number of electronic and social media methods for keeping track of what our subjects are eating. These include:

* Initially daily, or near daily contacts for the first week of each diet, then at least weekly contacts, and then at least monthly contacts.
* online data system that monitors food and activity (e.g., the USDA super tracker, myfitnesspal, etc).
* tweets or texts that ask the subjects to go to an elink and answer a few questions, e.g., did you eat grains today? The answers are downloaded to a database that can be compiled to reflect dietary compliance for each subject.

We will also develop a secure website so that participants from each group can discuss with others what problems and solutions they are using.

Last, we will also assess 24 hour urines for creatinine, sodium, and potassium at 0, 16 and 32 weeks. Both of these diets will be higher in potassium and lower in sodium than typical American diets. Although we expect our subjects will be motivated enough to follow these diets, from our previous studies we have found that some subjects were not honest about what they were eating, and this was reflected in the 24 hour urine excretion of potassium and sodium.

Assays:

Samples will be drawn at time 0; week 8; week 16; week 24 and week 32. We will collect serum, plasma and urine at all these timepoints for banking. The following tests will be performed at time (table 2):

1. CBC, Chemical profile; blood lipids; cardiovascular risk factors and inflammatory cytokines and adipokines (time 0, week 16, week 32): Electrolytes, liver function tests, fasting glucose, lipid panel and insulin levels will be measured by Quest labs. PAI-1 will be measured by a colorimetric assay (Chemicon, Temecula, CA). Homocysteine, fibrinogen, hsCRP and ICAM-1 will be assayed by the UCSF clinical laboratory using standard analytical methods. Commercial kits will be used to measure fasting serum non-esterified fatty acids (Wako Diagnostics kit ;Richmond Virginia); serum TNF-α , IL-6, adiponectin and leptin (Quantikine HS high sensitivity ELISA ;R & D Systems, Minneapolis, MN
2. Systemic oxidative stress (time 0, weeks 16, 32): we will measure 4 serum markers of oxidative stress; protein carbonyls (a product of protein oxidation), TBARS (a measurement of lipid peroxidation), TRAP (a measure of total antioxidant activity), and isoprostanes (formed from the peroxidation of arachidonic acid in lipoproteins and membranes). Blood samples will be drawn in the fasted state both at initial screening and after ALA treatment. Protein carbonyls, TBARS, and TRAP will be performed at UC Davis Clinical Laboratories employing standard techniques. Serum 8-isoprostane-F2α will be measured by KRONOS Science laboratory, Phoenix Arizona. We will also measure urine markers of oxidative stress before and after CRLA treatment. These will include 8-isoprostane-F2α, and 8-hydroxy guanosine (a marker of oxidized DNA). These urine assays will be performed KRONOS Science laboratory, Phoenix Arizona and Dr Jack Roberts, Vanderbilt University.
3. Telomere assessment. The length of telomeres, the DNA caps at the ends of chromosomes, is emerging as an indicator of stress-related biological aging: Data have implicated accelerated telomere shortening in the context of increased psychological stress and stress arousal [10, 11]Blood drawn by a licensed phlebotomist (4 mL for telomere assessment) at baseline (0 weeks) and 16-weeks will be assayed for telomere length. Samples will be frozen and transferred on dry ice to the Blackburn Laboratory at UCSF, located at 600 16th Street, San Francisco, California, by a laboratory technician. Assays will be completed according to the polymerase chain reaction (PCR) method..
4. 24 hr urine collections . collections as per clinical protocol. We will measure volume, Na, K, pH, creatinine and calcium

   Reproductive testing:

   Subjects will undergo assessment of 1)SHBG and androgen levels: total testosterone, androstenedione and DHEAS; 2) clinical hyperandrogenism: hirsutism by modified Ferriman-Gallwey and acne scores; 3) menstrual cyclicity (cycle interval and pattern); and 4) ovarian morphology (follicle count and ovarian volume).

   Androgen levels (times 0, weeks 16, 32): Two serum samples will be obtained 30 minutes apart.. Serum will be isolated and aliquoted for future analysis of androstenedione (A), testosterone (T), DHEAS, 17 hydroxyprogesterone (17-OHP) and SHBG.

   Clinical hyperandrogenism: The presence and extent of hirsutism will be determined using a modification of the Ferriman-Gallwey (FG) scoring method[12] while acne will be scored according to the American Academy of Dermatology .Subjects will be requested to avoid any mechanical treatment for hair removal for 4 weeks prior to the baseline visit and to list all such treatments that are utilized during the study and their frequency.

   Menstrual cyclicity: Menstrual frequency will be assessed as a menstrual frequency ratio as described by Elkind-Hirsch [13]so that menstrual events are normalized to the normal interval of 12 menses per year (MFR=1.0) or, for instance, those with 6 cycles per year would have an MFR of 0.5.

   Ovarian morphology: All subjects will undergo a transvaginal ultrasound (TVUS) to obtain an antral follicle count at baseline, 8 and 16 weeks. The study investigator will image both the left and right adnexal areas in two planes, and make measurements of the transverse, longitudinal, and anteroposterior diameters of each ovary using electronic calipers on a Shimadzu SDU-450XL machine with a variable 4-8 mHz vaginal transducer. The examination of each adnexa will ensure an adequate opportunity to locate the organs. Inability to locate adnexa in this age group is less than 1% (internal data). All echo-free structures in the ovaries will be regarded as follicles. Follicles with a mean diameter (of two dimensions) between 2 and 10 mm will be counted. Calculation of all follicles (2-10mm), as well as those 2- 5mm, will be possible as these numbers will be recorded separately. The total between the two ovaries (2- 10mm) will be considered the AFC. The volume of each ovary will be calculated by measuring the three perpendicular diameters and applying the formula for an ellipsoid: (L x H x W x π/6). Data will be entered directly onto scannable datasheets. Examination will also determine whether cysts/other abnormalities exist and provide images to document number and type of abnormalities. Clinical alerts will be generated for ovarian cysts of greater than 3cm diameter or solid adnexal masses of any size. Dr. Huddleston will be responsible for relaying information about clinical alerts to patients and physicians.
5. Body composition: Total body water (TBW) and extracellular water (ECW) volumes will be determined by bioimpedance spectroscopy (Intermed Inc, Melbourne Australia) at baseline, 16 and 32 weeks. Subjects will also be weighed at each visit. We will also do waist and hip measurements at baseline, 16 and 32 weeks .
6. Blood pressure (BP) and heart rate (HR): These will be measured at each visit in the morning after 10 minutes of rest in the sitting position using an automated oscillometric device (Dinamap, Critikon Inc) programmed to obtain 3 readings within 3 minutes, and then will calculate average daily pressure

j. Questionnaires: Participants will complete the following questionnaires per the schedule specified in Table 1. Questionnaires tap psychological experience, health and eating behavior, and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the study is restricted to reproductive age women with PCOS
* Chronic oligo/anovulation defined as an intermenstrual interval of >45 days and/or < 8 menstrual cycles/year and evidence of either hyperandrogenemia (elevation of total or free testosterone above the normal range for women) and/or clinical hyperandrogenism (hirsutism and/or acne)
* Age 18-40
* Agreeable to avoidance of pregnancy and to use barrier contraception for duration of study
* BMI between 18 to 40 kg/m2

Exclusion Criteria:

* Other abnormalities which might lead to anovulation: hyperprolactinemia, thyroid dysfunction and other causes of hyperandrogenemia including late onset congenital hyperplasia
* Evidence of diabetes based on a fasting glucose >126 mg/dl or OGTT
* Use of medications and/or supplements that influence either ovarian function or insulin sensitivity, within 2 months: including oral contraceptive pills, hormonal implants, anti-androgens, antipsychotics or antihypertensives metformin, glucocorticoids, and/or health food remedies other than multi-vitamins and calcium;
* Subjects who are on oral contraception, metformin, or nutritional supplements must agree to discontinue these drugs and undergo an 8 week washout period before the tests are performed
* Alcohol usage more than 7 drinks/week
* Hemoglobin < 10 grams
* Smokers
* Inability to understand the study goals and protocols and the consent form
* Any subject, who in the opinion of the investigators, does not qualify for the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
menstrual cycle frequency | 4 months
  questionnaires, ovarian ultrasound for volume

SECONDARY OUTCOMES:
insulin sensitivity | 4 months
  fasting glucose and insulin, 2 hour oral glucose tolerance tests

CONTACTS AND LOCATIONS:
Overall Officials: Heather Huddleston, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
would share only with participant, if asked by participant

DOCUMENTS (1):
  • Informed Consent Form (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02190097/ICF_000.pdf